CLINICAL TRIAL: NCT01657552
Title: A Phase I, Open-label, Three-Period, Single Sequence, Crossover Study Evaluating the Drug-Drug Interaction Between Eltrombopag and Boceprevir and Between Eltrombopag and Telaprevir in Healthy Adult Subjects
Brief Title: Eltrombopag/Boceprevir and Eltrombopag/Telaprevir Drug-Drug Interaction Study In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 116010
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Thrombocytopaenia
Keywords: Drug interaction; INCIVEK (telaprevir),; SB-497115 (eltrombopag); Pharmacokinetics; Thrombocytopenia; VICTRELIS (boceprevir)
MeSH Terms: conditions — Thrombocytopenia | interventions — eltrombopag; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Eltrombopag (Experimental): Subjects will receive single oral dose of eltrombopag 200 mg in Period 1 with moderate-fat, low-calcium meal.
  Interventions: Drug: Eltrombopag
- Boceprevir (Experimental): Subjects will receive boceprevir 800 mg orally every 8 hours (hrs) for 10 days in Period 2 with moderate-fat meals.
  Interventions: Drug: Boceprevir
- Telaprevir (Experimental): Subjects will receive telaprevir 750 mg orally every 8 hours hrs for 10 days in Period 2 with moderate-fat meals.
  Interventions: Drug: Telaprevir
- Eltrombopag and Broceprevir (Experimental): Subjects will receive eltrombopag 200 mg as single oral dose and boceprevir 800 mg orally every 8 hrs for a day in Period 3 with moderate-fat meals.
  Interventions: Drug: Eltrombopag; Drug: Boceprevir
- Eltrombopag and Telaprevir (Experimental): Subjects will receive eltrombopag 200 mg as single oral dose and telaprevir 750 mg orally every 8 hrs for a day in Period 3 with moderate-fat meals.
  Interventions: Drug: Eltrombopag; Drug: Telaprevir

INTERVENTIONS:
Drug: Eltrombopag — Each tablet contains 100 mg of Eltrombopag (Dose 200 mg)
  Arms: Eltrombopag; Eltrombopag and Broceprevir; Eltrombopag and Telaprevir
Drug: Boceprevir — Each capsule contains 200 mg of Boceprevir (Dose 800 mg)
  Arms: Boceprevir; Eltrombopag and Broceprevir
Drug: Telaprevir — Each tablet contains 375 mg of Telaprevir (Dose 750 mg)
  Arms: Eltrombopag and Telaprevir; Telaprevir

SUMMARY:
The purpose of the current Phase I, open-label, three-period, single sequence, crossover study, TPL116010, is to evaluate the potential drug-drug interaction between eltrombopag (ELT) and bocrprevir (BCP) and between ELT and telaprevir (TLP) in healthy subjects. In this study there will be a screening visit, three treatment periods, and a follow-up visit. In Period 1, subjects will receive a single dose of ELT on Day 1, and pharmacokinetic (PK) sampling will occur for 72 hours. In Period 2, subjects will receive BCP/TLP for 10 days with PK sampling for 8 hours. In Period 3, subjects will receive a single dose of ELT with BCP/TLP on Day 1 only with PK sampling for 72 hours. Subjects will return for a follow-up visit within 10 to 14 days of the last dose of study drugs. The total duration of the study from Screening to Follow-up will be approximately 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with no clinically significant abnormality identified by physician by evaluation of medical history, physical examination, clinical laboratory tests or electrocardiogram (ECG).
* Able to swallow and retain oral medication.
* Male or female subjects between the ages of 18 to 64 years of age inclusive, at the time of signing the informed consent.
* Capable of giving written informed consent which includes compliance with the requirements and restrictions listed in the consent form. Signed informed consent must be on file prior to screening procedures.
* Body weight >= 50 kilogram (kg) (110 pounds [lbs]) for men and >=45 kg (99 lbs) for women and body mass index (BMI) of 18.5 to 32.0 kg/ (meters squared) m^2 inclusive.
* Male subjects, who are not surgically sterile, must agree on abstinence or to use a double barrier method, such as, a condom plus spermicidal agent (foam/gel/film/cream/suppository). This criterion must be followed from the time of the first dose of study medication until 14 days after the last dose of medication.
* A female subject is eligible to participate if she is neither pregnant nor lactating, and falls into one of the following categories: non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or bilateral oophorectomy, or postmenopausal females defined as being amenorrheic for greater than 1 year and having serum estradiol and follicle stimulating hormone levels consistent with menopause, child-bearing potential with negative beta human chorionic gonadotropin (βhCG) test and agrees to comply with recognized non-hormonal contraceptive methods from screening or at least two weeks prior to first dose (whichever is earlier) until the follow-up visit. Recognized non-hormonal contraceptive methods include: complete abstinence from intercourse, two forms of barrier contraception (e.g. condom with spermicide, or diaphragm with spermicide), or intrauterine device (IUD).

Exclusion Criteria:

* History of Gilbert's syndrome.
* History of deep vein thrombosis or other thromboembolic event.
* History of thrombocytopenia or bleeding due to abnormal platelet number or function.
* Clotting factor abnormalities associated with hypercoagulability, including Factor V Leiden, Protein C or Protein S deficiency or antithrombin III deficiency.
* Elevated blood pressure (BP) at screening, Day -1 and at pre-dose (systolic >140 mm Hg [millimeters of mercury], diastolic >90 mmHg). If the subject's BP is elevated on the first measurement, complete two additional BP measurements at least 2 minutes apart and average the three assessments to evaluate this criterion. If averaged BP exceeds the safety criteria, the subject should be excluded.
* History of atrial fibrillation, mitral valve prolapse, significant heart murmur or vascular bruit.
* Prolonged QTcF interval at screening, Day 1 and at pre-dose (for females and males >450 milliseconds [ms]). If the QTcF interval is prolonged on the initial ECG, then complete two additional ECGs at least 5 minutes apart and take the average QTcF measurements of all three ECGs to evaluate this criterion. If averaged QTcF exceeds the safety criteria, the subject should be excluded.
* Female subjects currently receiving hormone replacement therapy (HRT).
* Positive for HIV, hepatitis B virus infection or HCV infection at screening.
* Positive urine drug screen including serum alcohol at screening or pre-dose (Day -1).
* History of alcohol/drug abuse or dependence within 12 months of the study. History of alcohol consumption in the past six months exceeding 7 units/week for women and 14 units/week for men (where 1 unit = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor).
* Urinary cotinine levels indicative of smoking at screening or pre-dose (Day -1). History of regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs (including aspirin and non-steroidal anti-inflammatory drugs [NSAIDs]), vitamins, herbal and dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer, such as St. John's Wort) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Subjects who have donated plasma within 7 days prior to the screening visit or where participation in this study would result in donation of blood in excess of 500 milliliters (mL) within a 56-day period.
* History of sensitivity to any of the study medications, or components thereof.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2012-10-26 (Actual); Study Completion 2012-10-26 (Actual)

PRIMARY OUTCOMES:
Composite pharmacokinetic (PK) parameters of eltrombopag following administration of boceprevir for 10 days with a single dose of eltrombopag | For 17 days
  Plasma eltrombopag PK Parameters: area under the concentration time-curves from time zero to infinity AUC(0-infinity) and maximum concentration (Cmax).
Composite PK parameters of boceprevir following administration of boceprevir for 10 days with a single dose of eltrombopag | For 17 days
  Plasma boceprevir PK Parameters: AUC from time zero to the dosing interval AUC(0-τ), Cmax, and Concentraction at end of the dosing interval (Cτ)
Composite PK parameters of eltrombopag following administration of telaprevir for 10 days with a single dose of eltrombopag | For 17 days
  Plasma eltrombopag PK Parameters: AUC(0-infinity) and Cmax
Composite PK parameters of telaprevir following administration of telaprevir for 10 days with a single dose of eltrombopag | For 17 days
  Plasma telaprevir PK Parameters: AUC(0-τ), Cmax, and Cτ.

SECONDARY OUTCOMES:
Composite PK parameters of eltrombopag following administration of boceprevir for 10 days with a single dose of eltrombopag | For 17 days
  Plasma eltrombopag PK Parameters: AUC from time zero to the last measurable concentration (AUC(0-t)), AUC obtained by extrapolation (%) (%AUCex), time from administration to first quantifiable concentration (tlag), time from administration to Cmax (tmax), elimination half life (t1/2), and apparent clearance (CL/F).
Composite PK parameters of boceprevir following administration of boceprevir for 10 days with a single dose of eltrombopag | For 17 days
  Plasma boceprevir PK Parameter: tmax.
Composite PK parameters of eltrombopag following administration of telaprevir for 10 days with a single dose of eltrombopag | For 17 days
  Plasma eltrombopag PK Parameters: AUC(0-t), %AUCex, tlag, tmax, t1/2, and CL/F.
Composite PK parameters of telaprevir following administration of telaprevir for 10 days with a single dose of eltrombopag | For 17 days
  Plasma telaprevir PK Parameter: tmax.
Safety and tolerability as assessed by the collection of adverse events | For 28 days
Safety and tolerability as assessed by change from baseline in clinical laboratory tests | For 28 days
  Clinical laboratory tests include hematology, clinical chemistry, urinalysis tests.
Safety and tolerability as assessed by change from baseline in vital sign | For 28 days
  Vital sign measurements will include systolic and diastolic blood pressure and pulse rate.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

REFERENCES:
- See also: Results for study 116010 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116010?search=study&study_ids=116010#rs